CLINICAL TRIAL: NCT05035524
Title: A Randomized Controlled Trial to Investigate The Role of Adjuvant Inhalable Sodium Bicarbonate Solution 8.4% in Treatment of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SB-COVID
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: COVID-19 Pneumonia; Covid19; COVID-19 Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19 | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Bicarbonate (Active Comparator): Adjuvant SB treatment Inhalation of SB 8.4% via a jet nebulizer (5 ml every 4 h) starting at 7:00 to 23:00 hours every day for 30 days together with instillation of SB 8.4% drops 4-times daily (three drops for each nostril) were offered to all patients in the study group
  Interventions: Drug: Sodium Bicarbonate Solution
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Bicarbonate Solution — Inhalation of SB 8.4% via a jet nebulizer (5 ml every 4 h) starting at 7:00 to 23:00 hours every day for 30 days together with instillation of SB 8.4% drops 4-times daily (three drops for each nostril) were offered to all patients in the study group (El-Badrawy et al., 2019).
  Other Names: Sodium Bicarbonate
  Arms: Sodium Bicarbonate
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate the role of SB 8.4% as adjuvant therapy in the treatment of COVID- 19 patients proved to be RT-PCR positive (mild, moderate and severe).

DETAILED DESCRIPTION:
Corona virus disease 19 (COVID-19) is a rapidly spreading disease that involves almost every part of the world. Although numerous attempts are being carried out to prevent and treat the disease, there is no consensus about the gold standard treatment. In the recent study (El-Badrawy et al., 2021) our group published a controlled study investigating the role of inhalable sodium bicarbonate (SB) as adjuvant treatment of non-severe CT- identified COVID-19 pneumonia. The study concluded that sodium bicarbonate 8.4% inhalation with its nasal instillation could be a possible adjuvant therapy for patients with non-severe COVID-19 pneumonia. Nevertheless, our previous study suffers from some limitations being non randomized, with a small sample size and short duration of follow up. Moreover, the study included only moderate cases of COVID-19 and excluded mild and severe cases.

The present protocol is designed to avoid the limitations of our previous study in an attempt to obtain clear answer about the role of inhalable SB as an adjuvant treatment of COVID-19.

The emergence of new mutants of Corona virus is a new problem that can face the synthesized new anti COVID vaccines. The use of SB in treatment of COVID-19 may overcome Corona virus whatever its mutant variant.

We hypothize that SB may neutralize the effect of sialic acid through change of pH and change of the negative change, therefore prevent attachment, fusion and transport of the virus into the host cell.

Theory:

SB inhalation may affect COVID-19 in respiratory tract through the following mechanism (Singh et al., 2020):

1. Alkalinisation of cell lysosomes; a mechanism similar to that of CQ and HCQ as reported by Singh et al 2020 that inhibit viral entry, transport and post-entry events.
2. Reaction with sialic acid on respiratory epithelial cells by buffering of the negative charge or change the pH of sialic acid that prevent entry of viruses into respiratory epithelial cells and/ or reinfection of the released viruses from the infected cells.

   Aim of the study:

   The aim of the study is to investigate the role of SB 8.4% as adjuvant therapy in the treatment of COVID- 19 patients proved to be RT-PCR positive (mild, moderate and severe).

   Patients and Methods Duration of the study: In the period between September 2021 and March 2022 Place of the study: Isolation department (for hospitalized cases) and COVID-19 surveillance clinic (for mild cases treated at home), Mansoura University hospitals.

   Patients

   Inclusion Criteria:

   In the period between September 2021 and March 2022, all consecutive patients suspected as COVID-19 presented to the respiratory evaluation zone and outpatient clinic of our university will be subjected to RT-PCR test for COVID. Patients proved to be RT-PCR positive will be included in the present study. The study will include all grades of the diseases.

   Exclusion Criteria:

   Children less than 18 years, pregnant ladies, those who will refuse enrollment or discontinue follow up.

   Study Design:

   This is a prospective randomized controlled trial (RCT) including two arms: control group receiving standard treatment as per the routine protocol of the Egyptian Ministry of Health (Masoud et al., 2020) according to the degree of the disease, and a study group receiving the standard treatment in addition to the adjuvant inhalable SB.

   Method of randomization: Eligible patients will be randomly assigned in a 1:1 ratio to receive either the standard treatment in addition to the adjuvant inhalable SB or standard treatment alone.

   The study is open-label. Methods

   Baseline assessment:

   Both groups were subjected to the following; full history, clinical examination, complete blood count, C- reactive protein, D dimer, liver function and kidney function tests. Radiological assessment with chest CT scan.

   Clinical, laboratory and radiological investigations were done at the time of diagnosis before start of treatment, after one week, one month, two months, and three months.

   Clinical assessment of the disease was defined according to World Health Organization (WHO, 2021 (table 1) Table 1: WHO Severity definitions (World Health Organization, 2021) Critical COVID-19 Defined by the criteria for acute respiratory distress syndrome (ARDS), sepsis, septic shock, or other conditions that would normally require the provision of life-sustaining therapies such as mechanical ventilation (invasive or non-invasive) or vasopressor therapy

   Severe COVID-19:

   Defined by any of:

   Oxygen saturation < 90% on room air. Respiratory rate > 30 breaths/min in adults. Signs of severe respiratory distress (accessory muscle use, inability to complete full sentences, central cyanosis, or presence of any other general danger signs.

   Moderate disease Adolescent with clinical signs of pneumonia (fever, cough, dyspnea, fast breathing) but no signs of severe pneumonia, including SpO2 ≥ 90% on room air Mild disease Symptomatic patients (fever, cough, fatigue, anorexia, myalgias, diarrhea, nausea, vomiting, anosmia or ageusia) PCR +ve for COVID-19 without evidence of viral pneumonia or hypoxia.

   Baseline investigations:

   The following laboratory studies will be done for all patients (Samprathi & Jayashree, 2021):
   * a complete blood count (CBC),
   * CRP.
   * serum creatinine, and liver function tests
   * D-dimer.

   Radiological assessment by CT:

   • CT images for each patient will be assessed for the following abnormalities: ground-glass opacity (GGO), consolidation, nodules, number of lung lobes affection, interlobular septal thickening and pleural effusion. In cases of GGO and consolidation, the severity of the lung affection is evaluated according to Bernheim et al. (2020), with each of the five lung lobes assessed and scored for the degree of involvement and classified as: score 0, no involvement (0% affected); 1, minimal (1-25%); 2, mild (26-50%); 3, moderate (51-75%); and 4, severe (76-100%). A total severity score is obtained by summing the five lobe scores, with a range between 0 and 20. A score of 1-5 is graded as 'minimal', 6-10 as 'mild', 11-15 as 'moderate' and 16-20 as 'severe.

   Standard Treatment:

   * For mild cases: If the patient is old age > 60 years, has uncontrolled diabetes or hypertension, active malignancy, obesity with BMI > 40 or more than 3 symptoms, the recommended treatment is ivermectin 6 mg daily or Favipiravir 1600 mg twice daily the first day then 600 mg twice daily for 5 days
   * For moderate cases… Anti-virals Immune-modulators Anti-coagulation Favipiravir 1600 mg twice daily the first day then 600 mg twice daily for 5 days Steroid (dexamethasone 6 mg or its oral equivalent) if patient has severe dyspnea or CT scan showing rapid deterioration or saturation < 93% Prophylactic anticoagulant if D-dimer between 500-1000 and therapeutic anti-coagulation if D-dimer > 1000 Remdesivir for high risk population with saturation < 92% (200 mg loading dose on day 1, followed by 100 mg daily for 5 days
   * For severe and critical cases…. Anti-virals Immune-modulators Anti-coagulation Remdesivir (200 mg loading dose on day 1, followed by 100 mg daily for 5 days Steroid (dexamethasone 6 mg or methylprednisolone 1 to 2 mg/kg/24 hours) Tocilizumab 4-8 mg/Kg/day for 2 doses 12 to 24 hours apart after failure of steroid therapy to improve the case for 24 hours Prophylactic anticoagulant if D-dimer between 500-1000 and therapeutic anti-coagulation if D-dimer > 1000 or if severe hypoxemia

   Adjuvant SB treatment:

   Inhalation of SB 8.4% via a jet nebulizer (5 ml every 4 h) starting at 7:00 to 23:00 hours every day for 30 days together with instillation of SB 8.4% drops 4-times daily (three drops for each nostril) were offered to all patients in the study group (El-Badrawy et al., 2019).

   Place of Treatment:

   Mild cases: home isolation Moderate cases without risk factors will be treated at home as per the protocol of the Egyptian Ministry of Health (Masoud et al., 2020), while moderate cases with risk factors (old age > 60 years, uncontrolled diabetes or hypertension, active malignancy, obesity with BMI > 40 or saturation < 92%), severe and critical cases will be treated at Isolation department, Mansoura University hospitals.

   Severe cases will be treated at Isolation department, Mansoura University hospitals.

   Outcome measures will include the following:

   I. Clinical outcomes:
   * The time to recovery defined as the first day, during the 28 days after enrollment, on which a patient met the criteria for category 1, 2, or 3 on the eight-category ordinal scale by Beigel et al., (2020):

     * Scale 1, not hospitalized and no limitations of activities;
     * Scale 2, not hospitalized, with limitation of activities, home oxygen requirement, or both;
     * Scale 3, hospitalized, not requiring supplemental oxygen and no longer requiring ongoing medical care (used if hospitalization was extended for infection-control or other nonmedical reasons);
     * Scale 4, hospitalized, not requiring supplemental oxygen but requiring ongoing medical care (related to Covid-19 or to other medical conditions);
     * Scale 5, hospitalized, requiring any supplemental oxygen;
     * Scale 6, hospitalized, requiring noninvasive ventilation or use of high-flow oxygen devices;
     * Scale 7, hospitalized, receiving invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); and
     * Scale 8, death.
   * Clinical status at days 7, 14 and 30.
   * Number of days with supplemental oxygen.
   * Number of days with noninvasive ventilation or high-flow oxygen.
   * Number of days with invasive ventilation.
   * The incidence of new oxygen use, of noninvasive ventilation or high-flow oxygen, and of invasive ventilation.
   * Number of days of hospitalization.
   * Mortality.

   II. Laboratory and Radiological Outcome Measures:

   • For all patients, a complete blood count (CBC), CRP and D-dimer at baseline, day 7, day 30.

   • Radiological assessment using CT chest at baseline, one week and one month later.

   Risk of COVID-19 infection transmission to health care workers from nebulizers as a method for aerosol generation:

   The British National Institute for Health and Care Excellence (NICE) advises that patients with suspected or confirmed COVID-19 may continue to use their nebulizer because the aerosols produced by them are generated from fluid within the nebulizer chamber that does not carry patient-derived viral particles. Indeed, if a particle in the aerosol comes into contact with contaminated mucous membrane, it ceases to be airborne and therefore will not be aerosolized. In any case, healthcare workers should use appropriate hand hygiene (wash hands and put on fresh gloves) when helping patients remove nebulizers and oxygen masks (British Thoracic Society, 2020).

   Practical advices (Cazzola et al., 2021):
   1. Pre-nebulization

      • Washing hands

      • Ensure the device is clean

      • Ensure adequate protection for health care workers and bystander hosts
   2. During nebulization • Separate room or negative pressure room (hospital/clinic); when possible, outside the house on a porch or patio or in a garage and in any case, near open windows or in areas of increased air circulation (home) • Mouth piece preferred over facemask
   3. Post-nebulization

      * Cleaning and disinfection of nebulizer
      * Cleaning of the surface and areas of nebulization

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients suspected as COVID-19 presented to the respiratory evaluation zone and outpatient clinic of our university will be subjected to RT-PCR test for COVID.
* Patients proved to be RT-PCR positive will be included in the present study.

Exclusion Criteria:

* pregnant ladies
* who will refuse enrollment or discontinue follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
The time interval to recovery defined as the first day | 1 months
  assessed by subtracting the day of recovery from the day of infection

CONTACTS AND LOCATIONS:
Overall Officials: Tamer El-Hadidy, Principal Investigator — Mansoura University Hospital - Chest Departement; Rehab Ahmad Elmorsey, Principal Investigator — Mansoura University Hospital - Chest Departement; Ibrahim Badr, Principal Investigator — Mansoura University Hospital - Chest Departement; Mohammed shehta, Principal Investigator — Mansoura University Hospital - Chest Departement; Adel El-Badrawy, Principal Investigator — Mansoura University Hospital - Chest Departement
Locations (1):
- Mansoura University Hospital - Chest Departement, Al Mansurah, DK, Egypt

REFERENCES:
- [Derived] El-Badrawy MK, Elmorsey RA, Elhosiny MM, Shehta M, El-Hadidy TA, Abdelwahab IE, El-Badrawy A, Shokeir AA. Efficacy and Safety of Nebulized Sodium Bicarbonate in Adults with COVID-19 (SODIC): A Randomized, Single-Center, Double-Blinded, Controlled Trial. Curr Ther Res Clin Exp. 2025 May 22;103:100801. doi: 10.1016/j.curtheres.2025.100801. eCollection 2025. PMID 40656233